CLINICAL TRIAL: NCT05604963
Title: Hemithyroidectomy or Total-Thyroidectomy in 'Low-risk' Thyroid Cancers
Acronym: HoT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/136591
Record Dates: First submitted 2022-07-22; First posted 2022-11-03 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Differentiated Thyroid Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Two-stage Completion Thyroidectomy (Active Comparator): Patients randomised to this arm will undergo a 2nd operation to remove the remaining thyroid lobe.
  Interventions: Procedure: Total Thyroidectomy
- Group 1: Surveillance (No Intervention): Patients randomised to this arm will have no 2nd surgery and proceed directly to follow-up visits.
- Group 2: Hemi-thyroidectomy (Experimental): Patients randomised to this arm will have a single HT operation to remove thyroid lobe with the tumour.
  Interventions: Procedure: Hemithyroidectomy
- Group 2: Total Thyroidectomy (Active Comparator): Patients randomised to this arm will have a single TT operation to remove the entire thyroid gland.
  Interventions: Procedure: Total Thyroidectomy

INTERVENTIONS:
Procedure: Total Thyroidectomy — Total Thyroidectomy - surgical removal of entire thyroid gland
  Arms: Group 1: Two-stage Completion Thyroidectomy; Group 2: Total Thyroidectomy
Procedure: Hemithyroidectomy — Hemithyroidectomy - surgical removal of partial thyroid gland
  Arms: Group 2: Hemi-thyroidectomy

SUMMARY:
This is a multi-centre, randomised, non-inferiority, phase III study in patients with low risk differentiated thyroid cancer.

Patients will be identified via oncology multidisciplinary team meetings. There will be two sources of patients in the trial, with the same histological diagnoses and prognosis (i.e. recurrence risk):

* Group 1: Patients who have already had a HT for thyroid problems and are then subsequently diagnosed with low risk DTC will be randomised 1:1 to undergo surveillance only OR a second operation to remove the rest of their thyroid gland (two-stage total thyroidectomy).
* Group 2: Patients diagnosed with low risk DTC using cytology (Thy5) but no surgery performed will be randomised 1:1 to have either a hemi-thyroidectomy OR a single-stage total thyroidectomy.

The overall aim of the trial is to determine whether hemithyroidectomy is an acceptable and cost-effective surgical procedure compared to total thyroidectomy in low risk thyroid cancer. Overall, 456 patients will be recruited to the trial. Patients will be initially be followed up post-surgery then 12 monthly for 6 years.

ELIGIBILITY:
Group 1 (HT already performed prior to diagnosis)

Inclusion criteria

• Aged 16 or over

Papillary thyroid cancer:

* pT1b-2 (≤4cm) irrespective of molecular genetic markers
* R0 resection (clinically excised but microscopic R1 resected tumours at discretion of the local MDT)
* cN0 or pN0, pNX & pN1a (≤5 foci, no extranodal spread)
* Confined to thyroid or minimal extrathyroidal extension
* No higher risk histological variants on morphology (small foci allowed at the discretion of the local MDT)
* No angioinvasion NB. PTC is still eligible where microscopic invasion of endothelial lined small capillary vascular spaces and lymphatic channels are present. It becomes ineligible in the rare instances when there is definite invasion of a larger vascular structure such as a vein with smooth muscle in its wall.
* Encapsulated FVPTC with capsular invasion only
* Micro-PTC (≤1cm)

  * multifocal
  * unifocal with pN1a (≤5 foci; no extranodal spread)

Follicular thyroid cancer (FTC), including oncocytic or Hürthle cell carcinoma:

* pT1b-2 (≤4cm) irrespective of molecular genetic markers

  - Minimally invasive, with capsular invasion +/- minimal (≤4 foci) vascular invasion (the latter is now called encapsulated angioinvasive and is at the discretion of the MDT)
* Confined to thyroid or minimal extrathyroidal extension

Exclusion criteria

* >4cm
* unifocal pT1a (≤1cm) PTC or FTC (unless pN1a as above)
* NIFTP (non-invasive follicular thyroid neoplasm with papillary-like nuclear features)
* Anaplastic, poorly differentiated or medullary thyroid carcinoma
* R2
* gross extrathyroidal extension
* pT4 or macroscopic tumour invasion of loco-regional tissues or structures
* pN1a with >5 foci or extranodal spread
* pN1b
* M1
* Aggressive PTC with any of the following features:

  * Widely invasive
  * Poorly differentiated
  * Anaplastic
  * predominance of Tall cell, Columnar cell, Hobnail, Diffuse sclerosing and other higher risk variants
* FTC, including oncocytic or Hürthle cell cancer with any of the following features:

  * Minimally invasive with extensive vascular invasion (now called encapsulated angioinvasive) (>4 foci)
  * Widely invasive
  * Poorly differentiated
  * Anaplastic

Group 2 (DTC on cytology or after core biopsy, who has not had prior thyroid surgery yet)

Inclusion criteria

* Aged 16 or over
* 'low risk' differentiated thyroid cancer confirmed by cytology or core biopsy.
* cT1b-2 irrespective of molecular genetic markers
* cN0
* Contralateral lobe without suspicious nodule(s) (U2, or U3/U4 with Thy2 on FNAC)

Exclusion criteria

• M1

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
3 Year Recurrence Rate | From surgery to any signs or symptoms of the cancer or death assessed up to a maximum of 3 years from surgery date
  (defined as thyroid cancer recurrence, metastatic disease or death from thyroid cancer (whichever occurs first))

SECONDARY OUTCOMES:
5 Year Recurrence Rate | From surgery to any signs or symptoms of the cancer or death assessed up to a maximum of 5 years from surgery date
  (defined as thyroid cancer recurrence, metastatic disease or death from thyroid cancer (whichever occurs first))
Anatomical Site of Recurrence | From surgery to confirmed recurrence assessed up to a maximum of 5 years from surgery date
  Location of recurrence
Risk of Loco-Regional Recurrence | From surgery to confirmed recurrence assessed up to a maximum of 5 years from surgery date
  (based on time to recurrence in the neck only)
Number of Additional Investigations and Procedures after Surgery | 2-4 weeks and 6, 18, 30, 42, 54, 66 and 78 months from date of surgery
  Number of further investigations/procedures related to the patient's thyroid surgery or thyroid cancer e.g. imaging, blood test, biopsy etc.
Type of Additional Investigations and Procedures after Surgery | 2-4 weeks and 6, 18, 30, 42, 54, 66 and 78 months from date of surgery
  Type of further investigations/procedures related to the patient's thyroid surgery or thyroid cancer e.g. imaging, blood test, biopsy etc.
Voice Function | Surgical complications and severity: From surgery date to discharge, 2-4 weeks, 6 months and 18 months from date of surgery; Voice Function: Post-randomisation/pre-surgery, 2-4 weeks and 6, 18, 30, 42, 54, 66 and 78 months from date of surgery.
  Measured using the Voice Handicap Index questionnaire (VHI-10); scores range from 0-40 with higher scores indicating greater voice-related handicap
Surgical complications and severity | Surgical complications and severity: From surgery date to discharge, 2-4 weeks, 6 months and 18 months from date of surgery; Voice Function: Post-randomisation/pre-surgery, 2-4 weeks and 6, 18, 30, 42, 54, 66 and 78 months from date of surgery.
  Using CTCAE v5.0 and the highest grade of each event type for each patient
Requirement for Hormone Replacement Therapy | From surgery date to discharge, 2-4 weeks and 6, 18, 30, 42, 54, 66 and 78 months from date of surgery.
  (percentage of patients who require this therapy compared between the trial arms)
Health Related Quality of Life | Baseline (post-randomisation/pre-surgery), 2-4 weeks and 6, 18, 30, 42, 54, 66 and 78 months from date of surgery.
  Measured using EORTC QLQ-C30; Scales range from 0-100 with higher scores for the functioning scales and global health status indicating higher QoL and higher scores on the symptom and single-item scales indicating lower QoL
Health Related Quality of Life | Baseline (post-randomisation/pre-surgery), 2-4 weeks and 6, 18, 30, 42, 54, 66 and 78 months from date of surgery.
  Measured using EORTC QLQ-THY35; Scales range from 0-100 with higher scores indicating higher QoL and lower scores indicating lower QoL
Health Related Quality of Life | Baseline (post-randomisation/pre-surgery), 2-4 weeks and 6, 18, 30, 42, 54, 66 and 78 months from date of surgery.
  Measured using EQ5D-5L; EQVAS score ranges from 0-100 with higher scores indicating higher QoL and lower scores indicating lower QoL; EQ-5D-5L index scores range from -0.224-1 with higher scores indicating higher QoL and lower scores indicating lower QoL
Health Related Quality of Life | Baseline (post-randomisation/pre-surgery), 2-4 weeks and 6, 18, 30, 42, 54, 66 and 78 months from date of surgery.
  Measured using FoP-Q-SF; scores range from 12-60 with higher scores indicating lower QoL and lower scores indicating higher QoL
Cost and Health Resource Use | a. Baseline, 2-4 weeks and 6, 18, 30, 42, 54, 66 & 78 months from date of surgery. b. From surgery date to discharge, 2-4 weeks and 6, 18, 30, 42, 54, 66 & 78 months from date of surgery. c/d. 6, 18, 30, 42, 54, 66 & 78 months from date of surgery
  Measured using EQ-5D-5L (generic QoL)
Cost and Health Resource Use | a. Baseline, 2-4 weeks and 6, 18, 30, 42, 54, 66 & 78 months from date of surgery. b. From surgery date to discharge, 2-4 weeks and 6, 18, 30, 42, 54, 66 & 78 months from date of surgery. c/d. 6, 18, 30, 42, 54, 66 & 78 months from date of surgery
  Measured using EORTC QLQ-C30 (cancer-specific QoL)
Cost and Health Resource Use | a. Baseline, 2-4 weeks and 6, 18, 30, 42, 54, 66 & 78 months from date of surgery. b. From surgery date to discharge, 2-4 weeks and 6, 18, 30, 42, 54, 66 & 78 months from date of surgery. c/d. 6, 18, 30, 42, 54, 66 & 78 months from date of surgery
  Measured using EORTC QLQ-THY34 (Cancer site specific QoL)
Secondary Care Health Resource Use | a. Baseline, 2-4 weeks and 6, 18, 30, 42, 54, 66 & 78 months from date of surgery. b. From surgery date to discharge, 2-4 weeks and 6, 18, 30, 42, 54, 66 & 78 months from date of surgery. c/d. 6, 18, 30, 42, 54, 66 & 78 months from date of surgery
  Collected using eCRFs and retrospectively for the study period from data in the Hospital Episodes Statistics linked to records in the NCRAS
Primary Care Health Resource Use | a. Baseline, 2-4 weeks and 6, 18, 30, 42, 54, 66 & 78 months from date of surgery. b. From surgery date to discharge, 2-4 weeks and 6, 18, 30, 42, 54, 66 & 78 months from date of surgery. c/d. 6, 18, 30, 42, 54, 66 & 78 months from date of surgery
  Collected using eCRFs (Review of Primary Care Visits)

CONTACTS AND LOCATIONS:
Locations (35):
- United Kingdom (35):
  - Leighton Hospital, Crewe, Cheshire
  - Aberdeen Royal Infirmary, Aberdeen
  - Royal United Hospital, Bath
  - Queen Elizabeth Hospital, Birmingham
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Colchester Hospital, Colchester
  - Royal Derby Hospital, Derby
  - Ninewells Hospital, Dundee
  - NHS Lothian, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Forth Valley Royal Hospital, Falkirk
  - Medway Maritime Hospital, Gillingham
  - NHS Greater Glasgow & Clyde, Glasgow
  - Ipswich Hospital, Ipswich
  - Leicester Royal Infirmary, Leicester
  - Liverpool University Hospitals, Liverpool
  - Guy's Hospital, London
  - Lister Hospital, London
  - Northwick Park Hospital, London
  - St George's Hospital, London
  - The Royal Marsden Hospitals, London
  - University College London Hospital, London
  - Luton and Dunstable University Hospital, Luton
  - Northampton General Hospital, Northampton
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Derriford Hospital, Plymouth
  - University Hospitals Dorset NHS Foundation Trust, Poole
  - Queen Alexandra Hospital, Portsmouth
  - Royal Berkshire Hospital, Reading
  - Glan Clwyd Hospital (Betsi Cadwaladr University Health Board), Rhyl
  - Sheffield Teaching Hospitals, Sheffield
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: No